CLINICAL TRIAL: NCT06368726
Title: Results of the Application of 80 Sessions of tDCS for 12 Months in Children Between 6 and 11 Years Old With Autism Spectrum Disorder With Rare Diseases, Genetic Problems or PANDAS
Brief Title: Result of tDCS in ASD Children With Comorbidities Like PANDAS, Rare Genetic Diseases or Autoimmune Disorders
Acronym: tDCS&ASD
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Spanish Foundation for Neurometrics Development (Other)
Collaborators: Fundacion para la Salud Materno Infantil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFND04042024
Record Dates: First submitted 2024-04-05; First posted 2024-04-16 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Attention; Visual Perceptual Weakness; Social Behavior; Fluency Disorder; EEG With Periodic Abnormalities
MeSH Terms: conditions — Social Behavior | interventions — Transcranial Direct Current Stimulation; Risperidone; Diet; Speech Therapy

STUDY DESIGN:
Intervention Model Description: Two groups of childs: 90 childs receive tDCS treatment and 90 traditional treatments with Risperidone educational training, speech therapy and visual training.
Who Masked: Investigator
Masking Description: Assessments regarding clinical recovery will be conducted by an assessor blind to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Traditional ASD approach (Active Comparator): The childs receive their tradicional interventions, Risperidone according to child's weight, diet, educational or speech therapies, pictographs.
  Interventions: Drug: Risperidone
- This group of childs will receive tDCS sessions (Experimental): This children receive 100 sessions during 12 monts in 4 groups of 25 sessions 2 per week of 30 minutes with a separation between them of at least 72 hours
  Interventions: Device: tDCS or Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: tDCS or Transcranial Direct Current Stimulation — We use weak currents applied over the child's scalp over 30 minutes twice a week during 100 days
  Other Names: tES Transcranial Electrical Stimulation
  Arms: This group of childs will receive tDCS sessions
Drug: Risperidone — Risperidone Risperidone according to child's weighs
  Other Names: Diet, educational or speech therapies, pictographs
  Arms: Traditional ASD approach

SUMMARY:
Results of the application of 100 sessions of tDCS for 12 months in children between 6 and 11 years old with autism spectrum disorder with rare diseases, genetic problems or PANDAS

DETAILED DESCRIPTION:
tDCS will be applied to 90 children diagnosed with ASD with Mu activity in one of their two temporal lobes and to another 90 children tDCS will not be applied but rather conventional treatments such as the Denver method, etc., in addition to collecting their electroencephalograms in eyes open condition, evoked potentials will be performed. with Mismatch Negativity paradigm to calculate the P300 wave every 25 sessions with a rest of 5-6 weeks between every 25 sessions and the changes in voltage and frequency of the EEG will be analysed using FFT & PSD, as well as the latencies and amplitudes of its P300 wave.

ELIGIBILITY:
Inclusion Criteria:

* Age between 7 and 15 years old
* Diagnosis: PDD, ASD or PANDAS
* Have genetic alterations with geneticist reports like: mutation, random mating between organisms, random fertilization or crossing over (or recombination) between chromatids of homologous chromosomes during meiosis.
* Natural birth without caesarean or complications
* Normal Pregnancy

Exclusion Criteria:

* Head Trauma
* Brain Injuries like meningitis or encephalitis, including SaRS, Herpes or MERS infections
* Epilepsy
* Rare Diseases with Auto-Immune Disease
* Rare diseases with Endocrinology problems
* Fever or Biochemical problems in the First Blood Test (First Visit)
* Vaccines Reactions

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
FFT | 12 months
  Change in Voltage for every frequency band
Power Density Spectrum Changes or PSD | 12 Months
  Amplitude of the PSD
ERP MMN changes | 12 months
  Changes in P300 wave amplitude
ERP MMN Changes | 12 Monts
  Changes in P300 wave latency

SECONDARY OUTCOMES:
Attention | 12 months
  Using ATTC scale average Scale
Social Skills | 12 months
  We used SSRS Scale Total Teacher Scale
Language | 12 months
  GhostBusters Res Spoken Language and Listening Average Score from 40 Cards
Visual Contact | 12 months
  P200 wave amplitude in occipital lobe

CONTACTS AND LOCATIONS:
Overall Officials: Jean Neville, MD, Study Director — New Remedies Ltd
Locations (1):
- New Remedies, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Moliadze V, Lyzhko E, Schmanke T, Andreas S, Freitag CM, Siniatchkin M. 1 mA cathodal tDCS shows excitatory effects in children and adolescents: Insights from TMS evoked N100 potential. Brain Res Bull. 2018 Jun;140:43-51. doi: 10.1016/j.brainresbull.2018.03.018. Epub 2018 Apr 3. PMID 29625151
- [Result] Moliadze V, Schmanke T, Andreas S, Lyzhko E, Freitag CM, Siniatchkin M. Stimulation intensities of transcranial direct current stimulation have to be adjusted in children and adolescents. Clin Neurophysiol. 2015 Jul;126(7):1392-9. doi: 10.1016/j.clinph.2014.10.142. Epub 2014 Oct 28. PMID 25468234
- [Result] Palm U, Segmiller FM, Epple AN, Freisleder FJ, Koutsouleris N, Schulte-Korne G, Padberg F. Transcranial direct current stimulation in children and adolescents: a comprehensive review. J Neural Transm (Vienna). 2016 Oct;123(10):1219-34. doi: 10.1007/s00702-016-1572-z. Epub 2016 May 12. PMID 27173384
- [Result] Buchanan DM, Amare S, Gaumond G, D'Angiulli A, Robaey P. Safety and Tolerability of tDCS across Different Ages, Sexes, Diagnoses, and Amperages: A Randomized Double-Blind Controlled Study. J Clin Med. 2023 Jun 28;12(13):4346. doi: 10.3390/jcm12134346. PMID 37445385
- [Result] Antal A, Luber B, Brem AK, Bikson M, Brunoni AR, Cohen Kadosh R, Dubljevic V, Fecteau S, Ferreri F, Floel A, Hallett M, Hamilton RH, Herrmann CS, Lavidor M, Loo C, Lustenberger C, Machado S, Miniussi C, Moliadze V, Nitsche MA, Rossi S, Rossini PM, Santarnecchi E, Seeck M, Thut G, Turi Z, Ugawa Y, Venkatasubramanian G, Wenderoth N, Wexler A, Ziemann U, Paulus W. Non-invasive brain stimulation and neuroenhancement. Clin Neurophysiol Pract. 2022 May 25;7:146-165. doi: 10.1016/j.cnp.2022.05.002. eCollection 2022. PMID 35734582
- [Result] Luckhardt C, Schutz M, Muhlherr A, Mossinger H, Boxhoorn S, Dempfle A, Salvador R, Ruffini G, Pereira HC, Castelo-Branco M, Latinus M, Bonnet-Brilhault F, Siemann J, Siniatchkin M, Ecker C, Freitag CM. Phase-IIa randomized, double-blind, sham-controlled, parallel group trial on anodal transcranial direct current stimulation (tDCS) over the left and right tempo-parietal junction in autism spectrum disorder-StimAT: study protocol for a clinical trial. Trials. 2021 Apr 6;22(1):248. doi: 10.1186/s13063-021-05172-1. PMID 33823927
- [Result] Rothenberger A, Heinrich H. Electrophysiology Echoes Brain Dynamics in Children and Adolescents With Tourette Syndrome-A Developmental Perspective. Front Neurol. 2021 Feb 15;12:587097. doi: 10.3389/fneur.2021.587097. eCollection 2021. PMID 33658971
- [Result] Buchanan DM, Bogdanowicz T, Khanna N, Lockman-Dufour G, Robaey P, D'Angiulli A. Systematic Review on the Safety and Tolerability of Transcranial Direct Current Stimulation in Children and Adolescents. Brain Sci. 2021 Feb 10;11(2):212. doi: 10.3390/brainsci11020212. PMID 33578648
- See also: Related Info — http://www.deepbrain.uk